CLINICAL TRIAL: NCT03160014
Title: Safety and Pharmacokinetics/Pharmacodynamics of SHR3824 in Patients With Hepatic Impairment (Single-Center, Open-label, Parallel-Group, Single-Dose Study)
Brief Title: Safety and Pharmacokinetics/Pharmacodynamics of SHR3824 in Patients With Hepatic Impairment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR3824-109
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2016-06

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — henagliflozin

ARMS (4):
- healthy volunteers (Experimental): Drug: SHR3824 20mg/day, oral tablet, single dose
  Interventions: Drug: SHR3824
- Mild Hepatic Impairment (Experimental): Drug: SHR3824 20mg/day, oral tablet, single dose
  Interventions: Drug: SHR3824
- Moderate Hepatic Impairment (Experimental): Drug: SHR3824 20mg/day, oral tablet, single dose
  Interventions: Drug: SHR3824
- Severe Hepatic Impairment (Experimental): Drug: SHR3824 20mg/day, oral tablet, single dose
  Interventions: Drug: SHR3824

INTERVENTIONS:
Drug: SHR3824 — Drug: SHR3824 20mg/day, oral tablet, single dose

SUMMARY:
Comparison of the pharmacokinetics/Pharmacodynamics of the SHR3824 in Patients With Mild, Moderate and Severe Hepatic Impairment Compared with Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 75 years (inclusive)
* Body mass index should be between 18 and 33 kg/m2 (inclusive) (ie, a measure of one's weight in relation to height)
* Liver damage due to viral hepatitis, alcoholic liver disease, autoimmune hepatitis, primary biliary cirrhosis of the liver (except for patients with drug-induced liver injury)

Exclusion Criteria:

* allergic to SGLT2 inhibitor analogues or any other similar structure;
* lactose intolerance history or lactose intolerance;
* Suspected or diagnosed as liver cancer or with other malignant tumors;
* Alcoholic liver, autoimmune liver disease, liver transplantation history

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The area under the plasma concentration-time curve (AUC) of SHR3824 | 72 hours after dosing
  AUC (a measure of the body's exposure to SHR3824) will be compared between normal hepatic function patients and mild or moderate or severe hepatic dysfunction patients
The maximum plasma concentration (Cmax) of SHR3824 | 72 hours after dosing
  Cmax (a measure of the body's exposure to SHR3824) will be compared between normal hepatic function patients and mild or moderate or severe hepatic dysfunction patients.

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | 72 hours after dosing
  The number of volunteers with adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- XiJing Hospital, XiAn, Shanxi, China